CLINICAL TRIAL: NCT05251636
Title: A Double-Masked, Multi-center, Active Controlled Safety and Efficacy Study of Adjunct Episcleral Brachytherapy for Polypoid Choroidal Vasculopathy
Brief Title: Adjunct Episcleral Brachytherapy for PCV
Acronym: KILAUEA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Salutaris Medical Devices, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMD-202101
Record Dates: First submitted 2022-02-11; First posted 2022-02-23 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Age-Related Macular Degeneration; Polypoid Choroidal Vasculopathy
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- ESB adjunct to IAI (Experimental): Single ESB treatment adjunct to intravitreal aflibercept injections (IAI)
  Interventions: Radiation: Episcleral Brachytherapy; Drug: Aflibercept Injection
- IAI monotherapy (Active Comparator): Intravitreal aflibercept injections (IAI)
  Interventions: Drug: Aflibercept Injection

INTERVENTIONS:
Radiation: Episcleral Brachytherapy — Minimally invasive, single fraction brachytherapy
  Arms: ESB adjunct to IAI
Drug: Aflibercept Injection — Standard of Care intravitreal aflibercept injection

SUMMARY:
This study is investigating the use of episcleral brachytherapy (ESB) adjunct to aflibercept compared to aflibercept monotherapy for the treatment of polyploid choroidal vasculopathy (PCV) in patients experiencing an inadequate response to anti-VEGF monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Active PCV due to nAMD
* Incomplete response to anti-VEGF
* Received at least 3 consecutive and sequential anti-VEGF injections (no missed treatments)
* Ability to undergo ESB intervention

Exclusion Criteria:

* Sub-retinal fibrosis
* Type I or Type II diabetes mellitus
* Previous therapeutic radiation to the head or neck that may have resulted in radiation dose to the retina
* Study eye with BCVA of worse than 20 ETDRS letters (20/400 Snellen)
* Fellow eye with worse BCVA than the study eye or other vision-threatening disease not eligible for treatment
* Receiving anti-VEGF therapy for any reason other than AMD

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) | 12 months

SECONDARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) | 24 months
Central Retinal Thickness | 12 and 24 months
Lesion size | 12 and 24 months

IPD SHARING:
Plan to Share IPD: Undecided